CLINICAL TRIAL: NCT02474862
Title: RCT of a Tailored Walking Program to Reduce Stress Among Pregnant Women
Brief Title: Healthy Expectations - a Program for Pregnant Women Experiencing Depressive Symptoms
Acronym: HE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: Brown University (Other); Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Cynthia Battle, Associate Professor (Research), Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01NR014540-01A1 (NIH)
Record Dates: First submitted 2015-06-11; First posted 2015-06-18 (Estimated); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Depressive Symptoms; Pregnancy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prenatal Walking Program (Experimental): The Prenatal Walking Program (PWP) is a gentle walking intervention tailored for pregnant women. The PWP intervention consists of 3 components: 1) biweekly session with a study interventionist; 2) the use of activity monitors to increase motivation and self-monitoring; 3) incentives to promote intervention adherence.
  Interventions: Behavioral: Prenatal Walking Program
- Postpartum Prep Program (Active Comparator): In the Postpartum Prep Program control condition (PPP) participants will attend individually education sessions matched in number and duration to the sessions in PWP. PPP involves providing health information particularly relevant to expectant mothers, including both maternal and newborn wellbeing.
  Interventions: Behavioral: Postpartum Prep Program

INTERVENTIONS:
Behavioral: Prenatal Walking Program — PWP is a gentle walking intervention tailored for pregnant women.
  Arms: Prenatal Walking Program
Behavioral: Postpartum Prep Program — PPP participants will attend individually education sessions matched in number and duration to the sessions in PWP. PPP involves providing health information particularly relevant to expectant mothers, including both maternal and newborn well being.
  Arms: Postpartum Prep Program

SUMMARY:
This study is a randomized control trial (RCT) evaluating a Prenatal Walking Program (PWP) in comparison to a Postpartum Prep Program (PPP) comparison group for pregnant women experiencing depressive symptoms. In addition to assessing changes in depressive symptoms, the investigators will examine other key maternal outcomes (maternal functioning, pain, anxiety, stress, fatigue), as well as infant outcomes including birth record data (gestation, weight, Apgar scores, etc) and careful, in-person assessment of infant neurobiological functioning at 30 days postpartum.

DETAILED DESCRIPTION:
Depressive symptoms are prevalent among pregnant women, and they are consistently linked with adverse outcomes for both women and infants, including higher rates of spontaneous abortion, preeclampsia, operative delivery, and postpartum depression. Additional risks to offspring include pre-term delivery, neonatal growth retardation, low birth weight, and delayed developmental milestones. In spite of these risks, the vast majority of affected women do not pursue any type of mental health treatment. Many women are reluctant to use antidepressants - or anything that could potentially harm the baby - prenatally. Because pregnant women have unique concerns regarding treatment acceptability, a critical need exists to develop interventions that are not only efficacious in reducing depressive symptoms, but are also viewed as acceptable by pregnant women.

Increased physical activity has numerous advantages as a strategy for improving mood during pregnancy, and prior research has shown that physical activity interventions can be effective in treating depressive symptoms in the general population. Physical activity interventions are also inexpensive, safe, and associated with a variety of positive health outcomes.

In spite of its potential as an acceptable and efficacious strategy for improving prenatal mood, few studies have evaluated physical activity as an intervention for pregnant women with depressive symptoms. Existing exercise programs that have been tested for reducing depressive symptoms in the general population are not likely to be appropriate or feasible for pregnant women. In light of this important gap, the investigators interdisciplinary team developed a gentle, 10-week, pedometer walking intervention tailored for pregnant women, the Prenatal Walking Program (PWP) and preliminarily evaluated PWP in an open trial, finding the intervention to be safe, feasible, and acceptable.

The current RCT will now evaluate PWP in comparison to a health education control comparison group tailored for perinatal women, called the Postpartum Prep Program (PPP). In addition to assessing changes in depressive symptoms, the investigators will examine other key maternal outcomes (maternal functioning, pain, anxiety, stress, fatigue), as well as infant outcomes including birth record data and in-person assessment of infant neurobiological functioning. Further, the investigators will examine evidence for potential behavioral, psychological, and biological mechanisms of action that mediate a possible treatment effect. Up to 152 pregnant women reporting elevated depressive symptoms during the current pregnancy will be enrolled and randomized into one of two groups, PWP or PPP, and will participate in blinded follow-up evaluations at multiple time-points throughout pregnancy and postpartum.

ELIGIBILITY:
Inclusion Criteria:

1. women aged 18 or over
2. 12-27 weeks gestation with a healthy singleton pregnancy
3. English-speaking
4. cleared by prenatal provider for moderate intensity exercise
5. experiencing moderate depressive symptom elevations at time of enrollment (QIDS-C; 8-20); (6) physically inactive or low-active at time of enrollment (mean < 90 minutes/week of moderate intensity exercise, over the last 3 months).

Exclusion Criteria:

1. recently started pharmacologic or psychosocial treatment for depressive symptoms within the past 4 weeks, or recently changed dose or treatment regimen in the past 4 weeks
2. current/recent acute suicidal symptoms
3. current substance use disorder
4. psychotic symptoms or cognitive impairment
5. current eating disorder
6. current or lifetime bipolar disorder, schizophrenia, or schizoaffective disorder.

   * Finally, while the following will not exclude participants from enrollment in the study, women meeting these two criteria will be excluded from participating in the blood draw component examining inflammatory markers:
7. current significant physical or neurological illness, ie., acute or chronic infectious, inflammatory or immune disorders
8. regular use of aspirin or non-steroidal anti-inflammatory drugs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2015-03-24 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Depression symptom severity | Change from baseline in depression severity at week 10
  The Quick Inventory of Depression Symptoms (QIDS) is the primary outcome measure and will be used to assess depression symptom severity.

SECONDARY OUTCOMES:
Physical activity level | Change from baseline in physical activity level at week 10
  Objective measurement using accelerometry and self-report
Anxiety | Change from baseline in anxiety level at week 10
  State Anxiety Scale
Perceived stress | Change from baseline in perceived stress at week 10
  Perceived Stress Scale -10
Health status - Inflammatory Biomarker 1 | Change from baseline in health status at week 10
  plasma interleukin-6 (IL-6)
Health status - Inflammatory Biomarker 2 | Change from baseline in health status at week 10
  plasma IL-1 beta (IL-1β)
Health status - Inflammatory Biomarker 3 | (CRP).Change from baseline in health status at week 10
  plasma tumor necrosis factor - alpha (TNF- α)
Health status - Inflammatory Biomarker 4 | Change from baseline in health status at week 10
  serum high sensitivity C-reactive protein (CRP).
Physical functioning | Change from baseline in physical functioing at week 10
  Patient Reported Outcomes Measurement Information System (PROMIS)- Short Form v1.0 - Phys. Function 10a
Physical Pain | Change from baseline in pain at week 10
  Patient Reported Outcomes Measurement Information System (PROMIS)- Pain Short Form v1.0
Fatigue | Change from baseline in fatigue at week 10
  Patient Reported Outcomes Measurement Information System (PROMIS)- Short Form v1.0 - Fatigue 8a Participant Version
Pregnancy discomfort | Change from baseline in pregnancy at week 10
  Maternal Physical Discomfort Scale
Quality of life and satisfaction | Change from baseline in quality of life at week 10
  Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form
Attachment to fetus/infant | Change from baseline in attachment to the fetus at week 10
  Maternal Antenatal Attachment Scale
Infant Outcome | 30-days postpartum
  This outcome will be based on a composite of measures relating to labor & delivery outcomes (e.g. gestational age) and infant neurobehavioral functioning (i.e., the Neonatal Intensive Care Unit Network Neurobehavioral Scale; NNNS).

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Battle, PhD, Principal Investigator — Butler Hospitl/Brown Unversity
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No